CLINICAL TRIAL: NCT07238829
Title: Analgesic Efficacy of Ultrasound-Guided Transversalis Fascia Plane Block Versus Surgical Wound Infiltration After Open Inguinal Hernia Surgery: A Randomized Controlled Trial
Brief Title: Transversalis Fascia Plane Block Versus Surgical Wound Infiltration for Postoperative Analgesia in Open Inguinal Hernia Repair
Acronym: TFPB-WIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Giresun Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Ilke Tamdogan, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INGHER2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Inguinal Hernia Unilateral; Postoperative Pain Management; Regional Anaesthesia; Transversalis Fascia Plane Block
Keywords: transversalis fascia plane block; regional anaesthesia; inguinal hernia; analgesia
MeSH Terms: conditions — Hernia, Inguinal; Agnosia

STUDY DESIGN:
Intervention Model Description: This study employs a parallel-group, randomized controlled design. Participants undergoing elective unilateral open inguinal hernia repair are randomized into one of two intervention arms. In one group, patients receive an ultrasound-guided Transversalis Fascia Plane Block (TFPB), while in the other group, local anesthetic is infiltrated into the surgical incision site. Both interventions are administered in a standardized manner, and all participants receive the same spinal anesthesia protocol and postoperative analgesia regimen. The investigators responsible for postoperative assessments are blinded to group allocation. Postoperative pain scores, opioid consumption, and secondary outcome measures are recorded at predefined time intervals to compare the analgesic effectiveness of the two techniques.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Transversalis Fascia Plane Block (TFPB) (Active Comparator): An ultrasound-guided Transversalis Fascia Plane Block will be performed by injecting a standardized volume and concentration of local anesthetic between the transversus abdominis muscle and the transversalis fascia. The block will be administered immediately after spinal anesthesia, prior to postoperative transfer. All other perioperative management and postoperative analgesia protocols will be identical to those in the comparison arm.
  Interventions: Procedure: Ultrasound-Guided Transversalis Fascia Plane Block (TFPB)
- Surgical Wound Infiltration (Active Comparator): At the end of surgery, the operating surgeon will infiltrate a standardized volume and concentration of local anesthetic into the relevant tissue layers of the surgical incision. The infiltration will be performed immediately after skin closure. Participants in this arm will receive the same spinal anesthesia and postoperative analgesia regimen as those in the TFPB group.
  Interventions: Procedure: Surgical Wound Infiltration

INTERVENTIONS:
Procedure: Ultrasound-Guided Transversalis Fascia Plane Block (TFPB) — An ultrasound-guided Transversalis Fascia Plane Block will be performed by injecting a standardized volume and concentration of local anesthetic between the transversus abdominis muscle and the transversalis fascia. The block will be administered immediately after spinal anesthesia, prior to postoperative transfer. All other perioperative management and postoperative analgesia protocols will be identical to those in the comparison arm.
  Arms: Ultrasound-Guided Transversalis Fascia Plane Block (TFPB)
Procedure: Surgical Wound Infiltration — At the end of surgery, the operating surgeon will infiltrate a standardized volume and concentration of local anesthetic into the relevant tissue layers of the surgical incision. The infiltration will be performed immediately after skin closure. Participants in this arm will receive the same spinal anesthesia and postoperative analgesia regimen as those in the TFPB group.
  Arms: Surgical Wound Infiltration

SUMMARY:
The purpose of this clinical trial is to evaluate whether two different analgesic techniques - ultrasound-guided Transversalis Fascia Plane Block (TFPB) and surgical wound infiltration - can improve postoperative pain control in adult patients undergoing open inguinal hernia repair.

The key questions that this study aims to answer are:

Does TFPB reduce total intravenous opioid consumption within the first 24 postoperative hours compared with wound infiltration?

Does TFPB improve postoperative pain scores at rest and during movement compared with wound infiltration?

Does TFPB improve patient satisfaction, reduce the need for rescue analgesics, and enhance overall postoperative recovery quality?

If there is a comparison group:

The investigators will compare the effects of TFPB with wound infiltration to determine whether either technique provides superior postoperative analgesia and reduces opioid requirements.

Participants will be asked to:

Undergo open inguinal hernia repair under spinal anesthesia.

Be randomly assigned to one of two groups:

TFPB Group: Receive an ultrasound-guided transversalis fascia plane block with local anesthetic.

Wound Infiltration Group: Receive local anesthetic infiltration performed by the surgeon along the incision line.

Postoperatively:

Report pain scores at defined intervals.

Receive standardized IV analgesia with documentation of opioid consumption.

Allow assessment of rescue analgesic requirement.

Be monitored for adverse events and recovery outcomes.

DETAILED DESCRIPTION:
worldwide. Inadequate analgesia in the early postoperative period may lead to delayed mobilization, prolonged hospital stay, and increased opioid consumption. Accordingly, current international guidelines recommend multimodal analgesia strategies and the use of regional anesthesia techniques when appropriate (1). Surgical wound infiltration is a frequently used component of multimodal analgesia in groin surgery; however, its effectiveness may vary depending on the timing of administration, technique, and the homogeneity of local anesthetic spread, and its duration of action is often limited. Recent clinical series continue to report significant postoperative pain and notable opioid requirements following primary unilateral open repair (1).

In recent years, ultrasound-guided fascial plane blocks have gained increasing attention due to their more predictable spread and potential to provide longer-lasting analgesia (2). The Transversalis Fascia Plane (TFP) block is a truncal block achieved by injecting local anesthetic between the transversus abdominis muscle and the transversalis fascia, thereby targeting the T12-L1 spinal nerves. This anatomical distribution provides a strong physiological rationale for its use in inguinal region surgery (3).

Several studies have demonstrated that the TFP block can reduce postoperative pain scores and rescue analgesic requirements in pediatric herniotomy and adult groin surgeries (4). However, randomized controlled trials directly comparing the TFP block with surgical wound infiltration in open inguinal hernia repair remain limited. Existing evidence partly stems from comparisons with other fascial plane blocks (e.g., Quadratus Lumborum [QL], Transversus Abdominis Plane [TAP] block) or from studies in different types of groin surgery, such as subinguinal varicocelectomy (5-7). Therefore, whether the TFP block provides a clinically meaningful advantage over wound infiltration in open inguinal hernia repair is a clinically relevant question that remains to be definitively answered.

This study aims to compare the contribution of the Transversalis Fascia Plane Block (TFPB) and surgical wound infiltration to postoperative analgesia in patients undergoing elective unilateral open inguinal hernia repair. The primary hypothesis is that TFPB will reduce cumulative rescue opioid consumption during the first 24 postoperative hours compared with wound infiltration. The secondary hypotheses are that TFPB will decrease postoperative pain scores, prolong the time to first rescue analgesia, and improve patient satisfaction without increasing the incidence of postoperative nausea and vomiting (PONV) or other adverse events.

articipants will be randomized into one of two intervention arms.

In the TFPB group, an ultrasound-guided transversalis fascia plane block will be performed in the postoperative period using a standardized volume and concentration of local anesthetic.

In the Wound Infiltration group, local anesthetic will be infiltrated by the surgeon into the relevant layers of the incision site at the end of the surgery.

All patients will receive a standardized spinal anesthesia protocol and a uniform postoperative analgesia regimen. Postoperative pain scores and opioid consumption will be recorded at predefined time intervals. The investigators responsible for postoperative assessments will remain blinded to group allocation throughout the study.

Primary outcome measure:

Total opioid consumption during the first 24 postoperative hours.

Secondary outcome measures:

NRS pain scores at rest and during coughing, the number of patients requiring rescue analgesia, the incidence of postoperative nausea and vomiting, block-related complications, and overall patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for elective unilateral open inguinal hernia repair
* Planned anesthesia: spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status I-II
* Able to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m²
* Known hypersensitivity to local anesthetics used in the study (e.g., bupivacaine) or to analgesic medications
* Coagulopathy
* Infection or hematoma at the planned block site
* Significant systemic disease (such as chronic kidney disease, hepatic failure, chronic obstructive pulmonary disease, etc.)
* History of chronic pain or long-term analgesic use
* Inability to use the patient-controlled analgesia system
* Presence of psychiatric disorders
* Refusal to participate in the study.
* Cases with a surgical duration shorter than 30 minutes or longer than 180 minutes were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption within the first 24 postoperative hours | 0-24 hours after surgery
  Cumulative amount of intravenous rescue opioid (e.g., tramadol or morphine equivalent dose) administered during the first 24 postoperative hours, recorded from the post-anesthesia care unit through postoperative hour 24.

CONTACTS AND LOCATIONS:
Overall Officials: İlke TAMDOGAN, Asst. Prof., Principal Investigator — Giresun University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No
ndividual participant data will not be shared.

REFERENCES:
- [Result] Lopez-Gonzalez JM, Lopez-Alvarez S, Jimenez Gomez BM, Arean Gonzalez I, Illodo Miramontes G, Padin Barreiro L. Ultrasound-guided transversalis fascia plane block versus anterior transversus abdominis plane block in outpatient inguinal hernia repair. Rev Esp Anestesiol Reanim. 2016 Nov;63(9):498-504. doi: 10.1016/j.redar.2016.02.005. Epub 2016 Apr 8. English, Spanish. PMID 27067036
- [Result] Celik EC, Ozbey I, Aydin ME, Yayik AM, Oral Ahiskalioglu E, Tor IH, Ahiskalioglu A. Efficacy of transversalis fascia plane block as a novel indication for varicocelectomy surgery: prospective randomized controlled study. BMC Anesthesiol. 2023 Feb 7;23(1):48. doi: 10.1186/s12871-023-02009-z. PMID 36750790
- [Result] Fouad AZ, Abdel-Aal IRM, Gadelrab MRMA, Mohammed HMES. Ultrasound-guided transversalis fascia plane block versus transmuscular quadratus lumborum block for post-operative analgesia in inguinal hernia repair. Korean J Pain. 2021 Apr 1;34(2):201-209. doi: 10.3344/kjp.2021.34.2.201. PMID 33785672
- [Result] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Result] Tran Q, Boezaart AP, Neal JM. Fascial plane blocks: the next leap. Reg Anesth Pain Med. 2021 Jul;46(7):568-569. doi: 10.1136/rapm-2020-101992. No abstract available. PMID 34145068